CLINICAL TRIAL: NCT01481324
Title: Measurement of Compliance in Clubfoot Bracing Via a Novel Pressure Sensor
Brief Title: Outcomes of Compliance With Brace Wear in Clubfoot
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Kosair Charities, Inc. (Other)
Responsible Party: Principal Investigator, Todd Milbrandt, Principal Investigator, Shriners Hospitals for Children
Other Study IDs: SHC-Lex-101
Record Dates: First submitted 2011-11-15; First posted 2011-11-29 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Clubfoot
Keywords: Clubfoot; Compliance; Brace wear
MeSH Terms: conditions — Clubfoot; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Functioning Pressure Sensor Group: This group will have a functioning pressure sensor placed on the foot ankle orthosis. The group will be blinded as to whether or not the sensor is functioning.
- Non-Functioning Pressure Sensor Group: This group will have a non-functioning pressure sensor (a placebo) placed on the foot ankle orthosis. The group will be blinded as to whether or not the sensor is functioning.
- No Sensor Group: This group will not have a pressure sensor placed on the foot ankle orthosis.

SUMMARY:
It has been shown that compliance with brace wear can significantly improve the treatment outcome of idiopathic clubfoot deformities. Noncompliance rates have been estimated to be around 30-41% with initial orthosis wear after successful treatment with serial castings. These studies have depended on family logs and not objective data. With the development of a monitoring device, this study hopes to examine: (1) actual patient compliance, (2) comparisons of actual wear time and assumed wear time and (3) the relationship of patient wear with clinical outcomes.

Hypothesis:

Actual patient compliance in foot abduction orthoses (FAO) wear is less than self-reported compliance and noncompliance is correlated to future surgeries.

DETAILED DESCRIPTION:
It is necessary that treatment teams avoid making any assumptions about patient compliance. This study will objectively measure brace wear-rate in patients with clubfoot that have already been prescribed a foot ankle orthosis. The use of a monitoring device will be able to give objective data on actual patient compliance with brace wear. It is hypothesized that objective compliance data will allow physicians to better assess the patient's therapy progress and outcome, troubleshoot problems or issues associated with barriers to brace wear, and better educate families confronted with having a child with clubfoot. Long term goals will then attempt to determine whether certain brace designs can increase wear time thus decreasing the rate of clubfoot recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral clubfoot
* Birth to 3 years of age
* Has been successfully treated with Ponseti casting protocol

Exclusion Criteria:

* Any other prior treatment for clubfoot
* Other existing diagnoses or conditions

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All clubfoot patients scheduled to be placed in a foot ankle orthosis (FAO)
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Milbrandt, MD, Principal Investigator — Shriners Hospital for Children
Locations (1):
- Shriners Hospital for Children, Lexington, Kentucky, United States

REFERENCES:
- [Background] Changulani M, Garg NK, Rajagopal TS, Bass A, Nayagam SN, Sampath J, Bruce CE. Treatment of idiopathic club foot using the Ponseti method. Initial experience. J Bone Joint Surg Br. 2006 Oct;88(10):1385-7. doi: 10.1302/0301-620X.88B10.17578. PMID 17012432
- [Background] Dobbs MB, Morcuende JA, Gurnett CA, Ponseti IV. Treatment of idiopathic clubfoot: an historical review. Iowa Orthop J. 2000;20:59-64. PMID 10934626
- [Background] Haft GF, Walker CG, Crawford HA. Early clubfoot recurrence after use of the Ponseti method in a New Zealand population. J Bone Joint Surg Am. 2007 Mar;89(3):487-93. doi: 10.2106/JBJS.F.00169. PMID 17332096
- [Background] Dobbs MB, Rudzki JR, Purcell DB, Walton T, Porter KR, Gurnett CA. Factors predictive of outcome after use of the Ponseti method for the treatment of idiopathic clubfeet. J Bone Joint Surg Am. 2004 Jan;86(1):22-7. doi: 10.2106/00004623-200401000-00005. PMID 14711941
- [Background] Thacker MM, Scher DM, Sala DA, van Bosse HJ, Feldman DS, Lehman WB. Use of the foot abduction orthosis following Ponseti casts: is it essential? J Pediatr Orthop. 2005 Mar-Apr;25(2):225-8. doi: 10.1097/01.bpo.0000150814.56790.f9. PMID 15718907

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functioning Pressure Sensor Group | Non-Functioning Pressure Sensor Group | No Sensor Group
Started | 21 | 24 | 22
Month 1-Wear Rate Data | 15 | 16 | 8
Month 2-Wear Rate Data | 9 | 13 | 7
Month 3-Wear Rate Data | 7 | 11 | 6
Completed | 21 | 22 | 20
Not Completed | 0 | 2 | 2
Not completed — Missing Data | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Number analyzed in each group
Groups:
- Total: Total of all reporting groups
Arm/Group | Functioning Pressure Sensor Group | Non-Functioning Pressure Sensor Group | No Sensor Group | Total
Number analyzed (Participants) | 21 | 22 | 20 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 22 | 20 | 63
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 16 | 16 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Wear Rate Percentage (Number of Hours Per Day Brace Was Worn Out of the Recommended 24 Hours)
Description: Number of hours per day in brace will be measured by pressure sensor at the end of month 1, month 2 and month 3. Parent report of brace wear will also be documented at each of these timepoints. Wear rate percentage will be calculated by dividing the number of hours of brace wear (either actual as measured by the sensor or reported by parent diary) by the recommended 24 hours.
Time Frame: 3 months
Measure: Mean (Full Range); unit: percentage of time worn
Arm/Group | Functioning Pressure Sensor Group | Non-Functioning Pressure Sensor Group | No Sensor Group
Number analyzed (Participants) | 21 | 22 | 20
percentage of time worn
  Month 1 Actual Wear Rate | 91.7 [72.7 to 97] | NA [NA to NA] — No sensor data available | NA [NA to NA] — No sensor data available
  Month 2 Actual Wear Rate | 86.8 [60.5 to 96.3] | NA [NA to NA] — No sensor data available | NA [NA to NA] — No sensor data available
  Month 3 Actual Wear Rate | 77.1 [52.6 to 95.8] | NA [NA to NA] — No sensor data available | NA [NA to NA] — No sensor data available
  Month 1 Reported Wear Rate | 94.9 [93.1 to 98.7] | 95.5 [91.8 to 98.7] | 94.8 [84.3 to 98.8]
  Month 2 Reported Wear Rate | 95.6 [92.3 to 99.4] | 95.8 [90.6 to 98.0] | 94.9 [86.9 to 97.3]
  Month 3 Reported Wear Rate | 94.8 [82.8 to 99.6] | 89.4 [36.7 to 97.7] | 94.2 [89.5 to 97.3]

ADVERSE EVENTS:
Arm/Group | Functioning Pressure Sensor Group | Non-Functioning Pressure Sensor Group | No Sensor Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 0/22

LIMITATIONS AND CAVEATS:
As shown in the monthly completion numbers, most families complied during the first month of treatment. After the first month, not only did the wear rates drop significantly, but also the number of subjects reporting sensor and diary data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No